CLINICAL TRIAL: NCT06387251
Title: A Decentralized Study to Assess the Effects of a 30 Day-wellness Program on Digestive Health, Weight and Overall Well-being
Brief Title: Assess the Effects of a 30 Day-wellness Program on Digestive Health, Weight and Overall Well-being
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peryam & Kroll Research Corporation (Other)
Collaborators: Alticor Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2023-11-437-0003
Record Dates: First submitted 2024-03-07; First posted 2024-04-29 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-03

CONDITIONS: Digestive Health
MeSH Terms: interventions — Health Promotion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Protein Powder (Other): Participants in Group A used the green powder supplement, probiotic supplement and protein Powder.
  Interventions: Other: 30 day wellness program
- All-in-one Meal Powder (Other): Participants in Group B used the green powder supplement, probiotic supplement and All-in-one Meal Powder.
  Interventions: Other: 30 day wellness program

INTERVENTIONS:
Other: 30 day wellness program — 30 days and will evaluate the effects of sponsor-designed 30-day wellness program consisting of 3 supplement and functional food products, recommended diet, physical activity, hydration and mindfulness activities.

SUMMARY:
The digestive system is a pivotal component of human health, playing a crucial role in the absorption of nutrients, elimination of waste, and even influencing mental well-being. Poor digestive health can significantly impact one's quality of life and overall well-being. Issues such as bloating, constipation, or imbalanced gut microbiome can affect one's overall well-being. Moreover, the gut-brain connection underscores how digestive health can affect mental well-being. The gut can contribute to serotonin and energy production thus influencing one's mood, energy levels and cognitive functions, affecting one's emotional stability. Additionally, inadequate nutrient absorption from an imbalanced digestive system may lead to suboptimal health, weakening the body and causing fatigue. Overall, maintaining good digestive health is crucial not only for physical comfort but also for normal metabolism, immune function, cognitive abilities, sleep and skin health, ultimately enhancing the overall quality of life. Products designed by the sponsor contains a blend of ingredients recognized for their potential benefits in promoting digestive health (including prebiotics, probiotics, postbiotics, plant-based extracts and plant-based protein). Furthermore, it is well established in the literature that diet, exercise, hydration and mindfulness all impact our gut health and overall well-being. Therefore, this scientific study seeks to validate the efficacy of the combination of products and life-style changes by assessing its impact on gut health and related health aspects like weight, metabolic health, fitness level, energy/fatigue levels, satiety/hunger, food cravings, cognitive abilities and overall well-being.

DETAILED DESCRIPTION:
This is a two-groups, virtual study where participants consume the green powder, probiotic and protein or meal replacement products and follow diet, hydration, physical activity and mindfulness activity regiment daily and provide feedback through the fitness tracker data, various questionnaires and measurement of basic biometrics over 30 days. The two-group design was chosen to obtain the data on the effects of the greens, probiotic products and protein vs a meal replacement food on a diverse group of participants. A virtual study ensures a broader reach and caters to the current trend of decentralized studies, which are more flexible and participant-centric. The choice of collecting daily fitness tracker data, spaced questionnaires and biometrics is to capture both immediate and cumulative effects of the products and the life-style regimen on the participants' health. A placebo has not been incorporated as it is not feasible to design a true placebo products that would taste and look indistinguishable from the intervention and placebo to the life-style regiment with a diet, physical activity, hydration, mindfulness activities are not feasible. The participants will be blinded to the sponsor name, brand name, and the exact products name.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female
2. Aged 20-65 years
3. Anyone willing to comply with study requirements
4. Anyone with no known allergies to the ingredients listed in the products
5. Generally healthy - do not live with any uncontrolled chronic disease - but looking to improve their general life-style and diet

Exclusion Criteria:

1. Women who are pregnant, breastfeeding, or attempting to conceive
2. Already follow a healthy plant-based diet and exercise regularly
3. Anyone with pre-existing chronic conditions that would prevent participants from adhering to the protocol, including oncological and psychiatric disorders
4. Individuals with a known history of severe diagnosed digestive disorders (e.g., Irritable Bowel Syndrome (IBS), Irritable Bowel Disease (IBD), Crohn's disease) or gastrointestinal-track surgeries
5. Planning to undergo an invasive medical procedure or GI surgery during the study period
6. Regular intake of medications that may interfere with the study or study product, including laxatives, sedatives, beta-blockers, anti-acids, etc.
7. Chronic smokers
8. Anyone with a history of substance abuse
9. Allergy to the products ingredients
10. Anyone with known severe allergic reactions that require an Epi-Pen
11. Anyone unwilling to follow the study protocol or unable to commit to the regiment for 28 days
12. Anyone currently participating or planning to participate other research study(s)
13. Regular consumption of probiotics, fiber, or digestive health supplements within 3 weeks of the study
14. People who participated in a weight loss or similar program within less than 3 months ago.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2024-01-29 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Bristol Stool Scale | Baseline, Day 16, Day 30
  To examine the effectiveness the products and program regiment on digestive health outcomes Endpoint: Reduction in digestive symptoms Type 1 - Separate hard lumps Type 2 - lumpy and sausage like Type 3 - A sausage shape with cracks in the surface Type 4 - like a smooth, soft sausage or snake Type 5 - Soft blobs with clear cut edges Type 6 - Mushy consistency with ragged edges Type 7 - Liquid consistency with no solid pieces N/A
Digestive symptom frequency questionnaire | Baseline, Day 16, Day 30
  To examine the effectiveness the products and program regiment on digestive health outcomes Endpoint: Reduction in digestive symptoms 0= never
  1. 1 day per month
  2. 2 to 3 days per month
  3. 1 day per week
  4. More than 1 day per week
  5. Every day

SECONDARY OUTCOMES:
Waist Circumference | Baseline and Day 30
  To examine the impact of the products and Program on Weight Loss and Abdominal Fat Endpoint: Weight loss, reduction in Waist Circumference
  Self-measured by participants
Improvements in sleep | Baseline, Day 16, Day 30
  To examine the impact of the products and program sleep Endpoint: Sleep Quality
  Fitness tracker measured sleep score PROMIS Sleep disturbances 4a
  1. very good
  2. good
  3. fair
  4. poor
  5. very poor
Improvements in stress | Baseline, Day 16, Day 30
  To examine the impact of the products and program stress Endpoint: Stress Quality
  Fitness tracker measured stress score PROMIS Sleep disturbances 4a
  1. very good
  2. good
  3. fair
  4. poor
  5. very poor
Fitness Level | days 3-30
  To examine the impact of the products and program on participants physical activity Endpoint: Fitness level
  Fitness tracker measured daily steps
Satiety Responsiveness and Hunger | Baseline, Day 16, Day 30
  To examine the impact of the products and program on satiety and hunger Endpoint: Satiety, hunger
  Satiety Responsiveness and Hunger Subscale
  1. Strongly disagree
  2. Disagree
  3. Neither agree or disagree
  4. Agree
  5. Strongly agree
Craving Intensity | Baseline, Day 16, Day 30
  To examine the impact of the products and program on sweet and rich food cravings Endpoint: sweet or rich food cravings
  Intensity of Cravings subscale
  1. none at all
  2. significantly less than usual
  3. slightly less than usual
  4. as usual
  5. slightly more than usual
  6. significantly more than usual
  7. more than ever
Cognitive Abilities | Baseline, Day 16, Day 30
  To examine the impact of the products and program on physical and psychological fatigue Endpoint: Cognitive Abilities
  PROMIS Cognitive Abilities 6a
  1. Not at all
  2. A little bit
  3. Somewhat
  4. Quite a bit
  5. Very much
Fatigue | Baseline, Day 16, Day 30
  To examine the impact of the products and program on physical and psychological fatigue Endpoint: Fatigue/Energy
  PROMIS Fatigue 6a
  1. Not at all
  2. A little bit
  3. Somewhat
  4. Quite a bit
  5. Very much
Skin Appearance | Baseline and Day 30
  To examine the impact of the products and program on general skin appearance Endpoint: General Health
  Skin Appearance Satisfaction
  1. = very dissatisfied
  2. = somewhat dissatisfied
  3. = neither satisfied nor dissatisfied
  4. = somewhat satisfied
  5. = very satisfied
General Health | Baseline and Day 30
  To examine the impact of the products and program on general health Endpoint: General Health
  SF-36 Questionnaire - General Health sub Scale
  1. - Excellent
  2. - Very good
  3. - Good
  4. - Fair
  5. - Poor
  1 = Definitely true 2 = Mostly true 3 = Don't know 4 = Mostly false 5 = Definitely False
Program Feedback | Day 30
  To collect Participants feedback on the products and Program Endpoint: Likeness & Suitability of such regiment for broader use
  Which programs.......enjoyment? Diet plan Staying active Exercise Hydration Mindfulness activities Products None of the above
  Which products......enjoyment? Green Powder Supplement Probiotic Supplement Protein Powder All in one Meal Powder None of the above
  RATE HOW LIKELY WOULD YOU
  1. Extremely Unlikely
  2. Highly Unlikely
  3. Very Unlikely
  4. Unlikely
  5. Neutral
  6. Somewhat Likely
  7. Likely
  8. Very likely
  9. Extremely likely
  RATE HOW LIKELY WOULD YOU
  1. Very Unlikely
  2. Unlikely
  3. Don't know
  4. Likely
  5. Very likely

CONTACTS AND LOCATIONS:
Overall Officials: George e Brown II, Principal Investigator — Peryam & Kroll Research Corporation
Locations (1):
- Wilkins Research, Chattanooga, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-12-11): https://cdn.clinicaltrials.gov/large-docs/51/NCT06387251/ICF_000.pdf